CLINICAL TRIAL: NCT00001749
Title: Treatment of Diamond Blackfan Anemia With Antithymocyte Globulin and Cyclosporine A
Brief Title: Medical Treatment for Diamond Blackfan Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 980144; 98-H-0144
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-07

CONDITIONS: Fanconi's Anemia; Hematologic Disease
Keywords: Immune Suppression; Erythroid Hypoplasia; Congenital Anemia; Reticulocytopenia; Diamond Blackfan Anemia
MeSH Terms: conditions — Fanconi Anemia; Hematologic Diseases; Anemia, Diamond-Blackfan | interventions — Antilymphocyte Serum; Cyclosporine

INTERVENTIONS:
Drug: Antithymocyte globulin
Drug: Cyclosporine

SUMMARY:
Diamond Blackfan anemia (DBA) is a condition in which the bone marrow is underdeveloped. DBA is considered a congenital disease, meaning patients are born with it. In DBA there is a lack of cells that give rise to red blood cells. The other elements produced in the bone marrow, such as white blood cells and platelets, are normal.

Standard treatments used for this disorder such as steroids and bone marrow transplants are associated with failure, relapse, side-effects, increased morbidity, and even death. Two drugs, antithymocyte globulin (ATG) and cyclosporin have been used to treat DBA, but have only provided occasional responses. No study has ever combined these two drugs for the treatment of DBA.

This study is designed to explore the combined use of ATG and cyclosporine as a rational approach to the treatment of DBA.

DETAILED DESCRIPTION:
Diamond Blackfan anemia (DBA) is a constitutional pure red cell aplasia of unknown etiology. There is laboratory evidence for an immune mechanism and most patients respond to corticosteroids. However the relapse and failure rate are high, and corticosteroids are associated with many short and long term side effects. Patients who do not respond or who do not tolerate corticosteriods require lifelong red blood cell transfusion and iron chelation therapy. Allogeneic bone marrow transplantation is an option for those with a related histocompatible donor, but this procedure is associated with high mortality and morbidity. Other therapies have been tried without general success. Occasional responses to either ATG or cyclosporine have been reported, but no study has used both ATG and cyclosporine. In other blood/bone marrow disorders of immune etiology these drugs have synergistic effects. We propose a Phase II study to explore the combined use of ATG and cyclosporine as a rational approach to the treatment of Diamond Blackfan anemia.

ELIGIBILITY:
INCLUSION CRITERIA:

Diagnosis of DBA as characterized by a hyporegenerative anemia presenting in early childhood with reticulocytopenia, and low or absent erythroid precursors in the bone marrow.

Transfusion-dependence due to steroid failure or intolerance of steroid side effects.

Ineligible for or declining an allogeneic transplant.

Ages 3 to 75.

EXCLUSION CRITERIA:

Serum creatinine greater than 2 times normal or a creatinine clearance less than 50% normal.

SGPT or SGOT greater than 5 times normal.

History of epilepsy (any seizures besides childhood febrile seizures).

Current pregnancy or unwillingness to take oral contraceptives if menstruating.

Positive diepoxybutane (DEB) test for Fanconi anemia.

HIV positivity.

Inability or unwillingness to sign an informed consent, either by the patient, or in the case of a minor, by the parent or guardian responsible for the patient.

Underlying organ failure and/or those with a Karnofsky performance status of less than 1.

Treatment with androgens, prednisone greater than 10 mg/day, growth factors, or other immunosuppressive therapies within one month of protocol entry.

Ongoing treatment with Beta-adrenergic blocking drugs.

Previous treatment with ATG and concurrent CSA. Previous treatment with either drug alone is acceptable if greater than one year prior to study entry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25
Dates: Start 1998-07; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Casadevall N, Croisille L, Auffray I, Tchernia G, Coulombel L. Age-related alterations in erythroid and granulopoietic progenitors in Diamond-Blackfan anaemia. Br J Haematol. 1994 Jun;87(2):369-75. doi: 10.1111/j.1365-2141.1994.tb04924.x. PMID 7524624
- [Background] Ball SE, McGuckin CP, Jenkins G, Gordon-Smith EC. Diamond-Blackfan anaemia in the U.K.: analysis of 80 cases from a 20-year birth cohort. Br J Haematol. 1996 Sep;94(4):645-53. doi: 10.1046/j.1365-2141.1996.d01-1839.x. PMID 8826887
- [Background] Halperin DS, Freedman MH. Diamond-blackfan anemia: etiology, pathophysiology, and treatment. Am J Pediatr Hematol Oncol. 1989 Winter;11(4):380-94. PMID 2694854